CLINICAL TRIAL: NCT00203944
Title: International Adoption and Stress Response Study
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 11685A
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Stress
Keywords: Adoption; Stress Response; Child Development
MeSH Terms: conditions — Fractures, Stress | interventions — Growth and Development

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- international adopted infants: international adoptees making their first visit to international adoption clinic
  Interventions: Behavioral: Behavioral, Development
- Control infants

INTERVENTIONS:
Behavioral: Behavioral, Development
  Groups: international adopted infants

SUMMARY:
This study aims to provide information about the emotional and physiological responses of post-institutionalized children in both a stressful situation (immunization) and a play situation.

DETAILED DESCRIPTION:
During the last decade, international adoptions have doubled in the United States. Because many of these infants and children have experienced institutionalization and poor caretaking before their adoption, international adoptees have special medical and emotional needs that must be met by both their parents and pediatricians. Currently, most clinical information about these children has focused on their physical health status so that protocols for evaluation and treatment can be established. Some systematic research has also focused on their overall developmental status including both cognitive and motor capabilities. These studies show that most of the children are developmentally delayed upon arrival to the U.S. Furthermore, follow-up studies have found international adoptees to score (on the average) significantly lower in cognitive functioning than their nonadopted peers even after spending substantial time in their adopting homes and falling mostly within the normal range. Not surprisingly, children's level of functioning at older ages is related to the length of time spent in institutional care.

These findings are consistent with an emerging literature on the lingering effects of early adversity on children's development. Potent adverse circumstances may include the unbuffered effects of poverty, experience in an institutional setting, physical or sexual abuse, and parental negligence Regardless of the source, children who are not protected from these disadvantageous situations demonstrate changes in their behavior as well as their biophysiological regulation.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than 1 year old
* Adopted infants
* Control group of non-adopted infants

Exclusion Criteria:

* Children greater than 1 year old

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants from international adoption clinic for adoptees and U of C pediatric follow-up clinic for controls
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2002-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Cortisol response levels | At clinic visit before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Larry Gray, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States